CLINICAL TRIAL: NCT03725917
Title: Efficacy of a Protocol of Intervention in Physiotherapy in the Prevention of Diabetic Foot Ulcers in Patients With Diabetic Neuropathy
Brief Title: Patients With Diabetic Neuropathy Who Receive Physiotherapy Treatment Will Have a Decrease in Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Guido Gomez Chiguano, Clinical Research, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V2.0_16.07.18
Record Dates: First submitted 2018-10-24; First posted 2018-10-31 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Foot Ulcer; Diabetic Neuropathy Peripheral
Keywords: Prevention; Physiotherapy; Diabetic Foot Ulcer; Exercise Therapy; Manual Therapy
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: All assessments will be made by an experienced Podiatrist, who will not have other functions in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The intervention will be a progressive physiotherapy protocol formed by therapeutic exercise and manual therapy
  Interventions: Other: Physiotherapy protocol
- Control Group (No Intervention): The control group will not receive physiotherapy treatment.

INTERVENTIONS:
Other: Physiotherapy protocol — The intervention will consist of a physiotherapy protocol twice a week for twelve weeks. The protocol will be done in three phases, constituting each month, a phase of the protocol. The first two phases will include therapeutic exercise of progressive difficulty and manual therapy, while the last phase will include only one week of manual therapy and therapeutic exercise, the last three weeks being composed only of therapeutic exercise
  Other Names: Physical therapy protocol
  Arms: Experimental Group

SUMMARY:
This study evaluates the effects of a physiotherapy protocol (manual therapy and exercise) in the prevention of diabetic foot ulcers in patients with diabetic neuropathy. A group of participants will receive a physiotherapy protocol added to their usual medical treatment and the other group will not receive physiotherapy treatment.

DETAILED DESCRIPTION:
Neuropathic diabetic patients present alterations in joint mobility, plantar pressures and ankle and foot function, characteristics related to the development of ulcers.

In previous studies, it has been observed that physiotherapy protocols have produced improvements in joint mobility, magnitude of plantar pressures, distribution of plantar pressures, and improved function in the ankle and foot.

A 12-week progressive physiotherapy protocol composed of manual therapy and exercise could produce changes in foot and ankle characteristics in diabetic neuropathic patients related to tissue damage, resulting in a reduction in ulcerations.

ELIGIBILITY:
Inclusion Criteria:

* Participants with diabetes mellitus type 1 or type 2
* Patients with diabetic neuropathy
* Patients with no previous history of ulcers
* Patients with no previous history of lower limb amputations

Exclusion Criteria:

* Patients with neurological or orthopedic problems that make walking difficult (spasticity, cerebral palsy, poliomyelitis, rheumatoid arthritis)
* Severe vascular complications (arterial or venous ulcers)
* Patients with critical ischemia
* Patient who need walking aids (canes, crutches, splints etc.)
* Patients with a history of neuropathy with different etiology from diabetes mellitus.
* Patients with peripheral nervous lesions (traumatic origin, associated with surgical procedures, compression of spinal roots, plexus palsy, herpes zoster, polyradiculopathy, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the integrity of the skin (Ulceration) | Clinical evaluation will be conducted at pre-treatment, post- treatment 12 weeks, post- treatment 24 weeks, post- treatment 36 weeks, post- treatment 48 weeks and post- treatment 60 weeks
  An ulcer is considered a full thickness wound below the ankle in a diabetic patient, regardless of duration, including gangrene and necrosis.
  The evaluator will review the patient's medical records on the day of the evaluations, in order to assess if there has been an ulceration in the periods between evaluations and also perform a foot exploration to assess if the ulcer is present on the day of measurement.
  The Wagner system assesses ulcer depth and the presence of osteomyelitis or gangrene using the following grades: grade 0 (pre- or post-ulcerative lesion), grade 1 (partial/full-thickness ulcer), grade 2 (probing to tendon or capsule), grade 3 (deep with osteitis), grade 4 (partial foot gangrene) and grade 5 (whole foot gangrene).

SECONDARY OUTCOMES:
Change in maximum plantar pressure | Clinical evaluation will be conducted at pre-treatment, post- treatment 12 weeks, post- treatment 24 weeks, post- treatment 36 weeks, post- treatment 48 weeks and post- treatment 60 weeks
  The maximum plantar pressure of 10 areas of foot support (medial heel, lateral heel, midfoot, plantar area of each of the heads of the metatarsals from first to fifth, first toe and support area of the middle fingers from second to fifth) will be obtained through the F-Scan® system, a computerized pedobarographic analysis system. To express the maximum plantar pressure the newton per centimeter (N/cm) will be used.
Change in joint mobility | Clinical evaluation will be conducted at pre-treatment, post- treatment 12 weeks, post- treatment 24 weeks, post- treatment 36 weeks, post- treatment 48 weeks and post- treatment 60 weeks
  The mobility of the tibiofibular-talar joint, subtalar joint and the first metatarsophalangeal joint, both in loading and unloading, will be measured by goniometer.
Change in foot function index | Clinical evaluation will be conducted at pre-treatment, post- treatment 12 weeks, post- treatment 24 weeks, post- treatment 36 weeks, post- treatment 48 weeks and post- treatment 60 weeks
  The foot function index will be measured by adapting the Foot Function Index (FFI) Questionnaire to Spanish. The FFI is a questionnaire in which the answers are about the experience of the participant's previous week.
  It consists of 23 items divided into 3 subscales: pain, disability and limitation of activity. For each item there is an visual analog scale with values from 0 to 10. If the respondents do not find the question appropriate, they can leave it blank. Once the questionnaire is completed, all the points are added and divided by the maximum score that can be achieved with the items that have been filled out. The result obtained from each subscale is multiplied by one hundred, and rounded if necessary, to obtain values between zero and one hundred, the higher the value, the worse the patient's condition will be. The total function is obtained by calculating the average of the 3 subscale
Change in neurological function of the foot | Clinical evaluation will be conducted at pre-treatment, post- treatment 12 weeks, post- treatment 24 weeks, post- treatment 36 weeks, post- treatment 48 weeks and post- treatment 60 weeks
  Neurological function of the foot will be assessed using the Neuropathy Disability Score (NDS) instrument. The neurological function of the foot will be assessed using the NDS instrument. This allows the global assessment of neuropathy, by evaluating both long nerve fibers, which intervene in reflexes and vibratory sensitivity; as short fibers, involved in sensitivity to pain and temperature. It consists of a standardized examination of ankle reflexes and the perception of some sensory tests: pain, temperature and vibration. The minimum score of the NDS is 0 and the maximum score is 10, 5 in each leg. A score of 10 points indicates the complete loss of sensitivity and the absence of tendon reflexes. An NDS score ≥ 6/10 has a 2.3 times higher risk of developing a new ulcer in a 2-year follow-up period than those with a score of ≤ 5/10
Change in confidence in the balance for specific activities | Clinical evaluation will be conducted at pre-treatment, post- treatment 12 weeks, post- treatment 24 weeks, post- treatment 36 weeks, post- treatment 48 weeks and post- treatment 60 weeks
  Confidence and balance in specific activities will be assessed by adapting the ´´Activities Specific Balance Confidence Scale (ABC)'' to Spanish.
  The ABC scale is a 16-item questionnaire that assesses the level of confidence when performing a specific task without losing balance or becoming unstable. The score of each item varies between 0% (No confidence) and 100% (Total confidence). The final score is obtained by adding the value of each item, and dividing it by 16
Changes in the integral pressure-time | Clinical evaluation will be conducted at pre-treatment, post- treatment 12 weeks, post- treatment 24 weeks, post- treatment 36 weeks, post- treatment 48 weeks and post- treatment 60 weeks
  The integral pressure-time of 10 areas of foot support (medial heel, lateral heel, midfoot, plantar area of each of the heads of the metatarsals from first to fifth, first toe and support area of the middle fingers from second to fifth) will be obtained through the F-Scan® system, a computerized pedobarographic analysis system. To express the integral pressure-time the newton second per centimenter will be used (N.S/cm).

CONTACTS AND LOCATIONS:
Overall Officials: José L Lázaro Martínez, Study Director — Universidad Complutense de Madrid
Locations (1):
- Universidad Complutense de Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Background] Goldsmith JR, Lidtke RH, Shott S. The effects of range-of-motion therapy on the plantar pressures of patients with diabetes mellitus. J Am Podiatr Med Assoc. 2002 Oct;92(9):483-90. doi: 10.7547/87507315-92-9-483. PMID 12381797
- [Background] Cerrahoglu L, Kosan U, Sirin TC, Ulusoy A. Range of Motion and Plantar Pressure Evaluation for the Effects of Self-Care Foot Exercises on Diabetic Patients with and Without Neuropathy. J Am Podiatr Med Assoc. 2016 May;106(3):189-200. doi: 10.7547/14-095. PMID 27269974
- [Background] Sartor CD, Hasue RH, Cacciari LP, Butugan MK, Watari R, Passaro AC, Giacomozzi C, Sacco IC. Effects of strengthening, stretching and functional training on foot function in patients with diabetic neuropathy: results of a randomized controlled trial. BMC Musculoskelet Disord. 2014 Apr 27;15:137. doi: 10.1186/1471-2474-15-137. PMID 24767584
- [Background] Dijs HM, Roofthooft JM, Driessens MF, De Bock PG, Jacobs C, Van Acker KL. Effect of physical therapy on limited joint mobility in the diabetic foot. A pilot study. J Am Podiatr Med Assoc. 2000 Mar;90(3):126-32. doi: 10.7547/87507315-90-3-126. PMID 10740995